CLINICAL TRIAL: NCT01257165
Title: Driving Simulator Performance Related to Serum Concentrations of the Benzodiazepine-like Hypnotic Zopiclone
Brief Title: Driving Simulator Performance After Intake of Zopiclone Sleeping Pills
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: SINTEF Health Research (Other); Norwegian University of Science and Technology (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 60R020.05
Record Dates: First submitted 2010-11-29; First posted 2010-12-09 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Automobile Driving
Keywords: Automobile driving; Zopiclone; Drug safety; Traffic accidents
MeSH Terms: interventions — zopiclone; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Zopiclone 5 mg (Experimental): Zopiclone 5 mg pill + placebo pill + placebo drink
  Interventions: Drug: Zopiclone; Drug: Placebo pill; Drug: Placebo drink
- Zopiclone 10 mg (Experimental): 2 x zopiclone 5 mg pills + placebo drink
  Interventions: Drug: Zopiclone; Drug: Placebo drink
- Ethanol 0.8 g/L (Active Comparator): 2 x placebo pills + ethanol 50 g/70 kg
  Interventions: Drug: Ethanol; Drug: Placebo pill
- Placebo (Placebo Comparator): 2 x placebo pills + placebo drink
  Interventions: Drug: Placebo pill; Drug: Placebo drink

INTERVENTIONS:
Drug: Zopiclone — Zopiclone pill 5 or 10 mg, given orally as a single dose.
  Other Names: Imovane; Zopiklon; Zopiclon
  Arms: Zopiclone 10 mg; Zopiclone 5 mg
Drug: Ethanol — 50 mg per 70 kg body weight, given orally as a single dose
  Other Names: Alcohol; Ethyl alcohol
  Arms: Ethanol 0.8 g/L
Drug: Placebo pill — Placebo pill identical to zopiclone pill, given orally as a single dose
  Arms: Ethanol 0.8 g/L; Placebo; Zopiclone 5 mg
Drug: Placebo drink — Placebo drink, given orally as a single dose
  Arms: Placebo; Zopiclone 10 mg; Zopiclone 5 mg

SUMMARY:
Zopiclone, a widely used hypnotic drug, is frequently found in blood samples taken from drivers suspected of driving under the influence. In this study, the investigators aim to correlate zopiclone serum concentrations with degrees of driving impairment in healthy volunteers by use of a validated driving simulator. The investigators also aim to compare their results with the results from a previous study that investigated zopiclone impairment of cognitive and psychometric tests.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Caucasian ethnicity
* Age 25-35 years
* Possession of a driver's licence for at least five years

Exclusion Criteria:

* Score ≥ 2 on the modified Apfel-scale to assess risk for motion sickness(*)
* History of driving under the influence of alcohol and/or illicit substances
* History or presence of alcohol or illicit drug abuse
* Former abnormal reaction to any hypnotic drug
* History of strong averse reactions to blood sampling procedures
* Regular (daily) intake of any prescribed drug, or intake of grapefruit juice or herbal remedies that can influence the metabolism of zopiclone (e.g. St John's wort)
* History of severe allergic reactions, or significant mental, cardiovascular, renal or hepatic disorder, or other significant disease as judged by the investigators
* Detection of any drugs of abuse on pre-session urine drug screening

(*)Modified Apfel-criteria for prediction of postoperative nausea/vomiting:

1. Smoker? yes 0, no 1
2. History of nausea and/or vomiting following surgery, dental treatment, injections or similar procedures? yes 0, no 1
3. History of car sickness after 10 years of age? yes 0, no 1

A score of two or more points excludes participation.

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Standard deviation of lateral position (SDLP) on road | 1 h after intake of study medication (during a 30 min driving simulator test session)
  SDLP is a measure that quantifies the extent of car weaving while driving. It has been shown to correlate well with blood alcohol concentrations, and traffic accident risk.
Standard deviation of lateral position (SDLP) on road | 3,5 hrs after intake of study medication (during a 30 min driving simulator test session)
  SDLP is a measure that quantifies the extent of car weaving while driving. It has been shown to correlate well with blood alcohol concentrations, and traffic accident risk
Standard deviation of lateral position (SDLP) on road | 6,5 hrs after intake of study medication (during a 30 min driving simulator test session)
  SDLP is a measure that quantifies the extent of car weaving while driving. It has been shown to correlate well with blood alcohol concentrations, and traffic accident risk

SECONDARY OUTCOMES:
Average speed | 1 h, 3,5 hrs and 6,5 hrs after intake of study medication (during a 30 min driving simulator test session)
Standard deviation of speed | 1 h, 3,5 hrs and 6,5 hrs after intake of study medication (during a 30 min driving simulator test session)
Frequency of brake pedal pressures | 1 h, 3,5 hrs and 6,5 hrs after intake of study medication (during a 30 min driving simulator test session)
Frequency of accelerator pedal pressures | 1 h, 3,5 hrs and 6,5 hrs after intake of study medication (during a 30 min driving simulator test session)
Steering wheel movement speed and reversal frequency | 1 h, 3,5 hrs and 6,5 hrs after intake of study medication (during a 30 min driving simulator test session)
Driving behavior at incidents | 1 h, 3,5 hrs and 6,5 hrs after intake of study medication (during a 30 min driving simulator test session)
Clinical test for impairment (CTI) | 1,5 hrs, 4 hrs and 7 hrs after intake of study medication (after driving simulator test sessions)
  The Norwegian CTI is a 25-item clinical test that is administered by physicians on subjects suspected of driving under the influence of drugs. The test conclusion is either "impaired" or "not impaired".

CONTACTS AND LOCATIONS:
Overall Officials: Lars J Slørdal, MD, PhD, Principal Investigator — Norwegian University of Science and Technology